CLINICAL TRIAL: NCT06298825
Title: Effect of Sarcopenia on Prognosis of Patients With Acute Decompensated Heart Failure: a Prospective, Multi-center, Observational Cohort Study
Brief Title: S-ADHF：Sarcopenia in Patients With ADHF
Acronym: S-ADHF
Status: Not yet recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Huan Ma, Deputy Director of Cardiology, Director of the Department of Cardiac Rehabilitation, Guangdong Provincial People's Hospital
Other Study IDs: KY2024-148
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-01

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acute decompensated heart failure; Sarcopenia; prognosis; mortality; Kansas City Cardiomyopathy Questionnaire (KCCQ)
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sarcopenia: Acute decompensated heart failure with sarcopenia. Sarcopenia will be defined using the Asian Working Group for Sarcopenia (AWGS) criteria in the study. According to the guidelines, we can define participants as having sarcopenia when low muscle strength or physical performance coexisted with low skeletal muscle mass. We will define low muscle strength as handgrip strength <26kg for men and <18 kg for women, low physical performance as a walk speed of <1.0m/s for both sexes. We can use bioelectrical impedance analysis to measure the appendicular skeletal muscle mass. The appendicular skeletal muscle mass index (ASMI) is calculated as the sum of muscle mass in the extremities divided by the height squared (kg/m2). The cut-off values of <7.00 kg/m2 for men and <5.70 kg/m2 for women will be used.
- Non-sarcopenia: Acute decompensated heart failure without sarcopenia

SUMMARY:
This is a prospective, multi-center, investigator-initiated observational cohort study. Enrollment with a minimum of of 195 cases each for patients with and without sarcopenia. Each patient is followed up for 6 month, 1 year, 2 years or until the occurrence of death.This study will examine the correlation between sarcopenia and prognosis in different subgroups of patients, and explore the additive effect of different comorbidities and sarcopenia on prognosis in patients with acute decompensated heart failure.

DETAILED DESCRIPTION:
Guangdong Provincial People's Hospital will be the lead center, with an additional 4 hospitals designated as satellite centers for the study. Enrollment of up to 500 participants adults aged over 18 years hospitalized for ADHF is planned, with a minimum of of 195 cases each for patients with and without sarcopenia The sympathetic nervous activity, psychosocial factors, quality of life, physical function and baseline physical activity will also be observed and recorded at baseline. Each patient is followed up for 6 month, 1 year, 2 years or until the occurrence of death. The primary clinical outcome is all-cause mortality at 6 months. Other clinical outcomes of interest include cardiovascular mortality, all-cause hospitalisation, HF hospitalisation, the frequency and length of hospitalization of patient readmitted and survival time from enrollment to death of deceased patients.

This study will examine the correlation between sarcopenia and prognosis in different subgroups of patients, and explore the additive effect of different comorbidities and sarcopenia on prognosis in patients with acute decompensated heart failure. S-ADHF will provide important information and evidence on the clinical aspects of sarcopenia in patients with ADHF, and will potentially and contribute to accurate risk stratification and optimal clinical management for patient with ADHF.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. At least one symptom of heart failure upon admission:Dyspnea at rest or with exertion, orthopnea, paroxysmal nocturnal dyspnea or exertional fatigue.
3. At least two of the signs of heart failure (HF):

Distended jugular veins, enlarged cardiac silhouette, apex beat displacement, third heart sound, or increased jugular venous pressure/central venous pressure/pulmonary capillary wedge pressure.

Pulmonary edema or pulmonary congestion (rales or chest X-ray/CT evidence of pulmonary congestion).

Peripheral edema. Elevated B-type natriuretic peptide (>100 pg/ml) or elevated N-Terminal Pro-Brain Natriuretic Peptide (>300 pg/ml).

Willingness to provide informed consent and cooperate with the follow-up

Exclusion Criteria:

1. Unable to understand and comply with protocol or to give informed consent
2. End-stage diseases other than heart failure, life expectancy <1 year, such as malignant tumors
3. Current or planned participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment of up to 500 participants adults aged over 18 years hospitalized for ADHF is planned, with a minmum of of 195 cases each for patients with and without sarcopenia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 6 months
  Number of all-cause death 6 months from hospital discharge

SECONDARY OUTCOMES:
All-cause mortality | 1 year and 2 year
  Number of all-cause death 1year and 2 years from hospital discharge
Cardiovascular mortality | 6 moths， 1year and 2 years
  Number of cardiovascular death 6 moths， 1year and 2 years from hospital discharge
All-cause hospitalisation | 6 moths， 1year and 2 years
  Number of all-cause hospitalisation 6 moths， 1year and 2 years from hospital discharge
HF hospitalisation | 6 moths， 1year and 2 years
  Number of HF hospitalisation 6 moths， 1year and 2 years from hospital discharge

OTHER OUTCOMES:
The frequency and length of hospitalization of patient readmitted | 6 moths， 1year and 2 years
  The frequency and length of hospitalization of patient readmitted
Survival time from enrollment to death of deceased patients | 6 moths， 1year and 2 years
  Survival time from enrollment to death of deceased patients

CONTACTS AND LOCATIONS:
Locations (1):
- Huan Ma, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savarese G, Lund LH. Global Public Health Burden of Heart Failure. Card Fail Rev. 2017 Apr;3(1):7-11. doi: 10.15420/cfr.2016:25:2. PMID 28785469
- [Background] Arrigo M, Jessup M, Mullens W, Reza N, Shah AM, Sliwa K, Mebazaa A. Acute heart failure. Nat Rev Dis Primers. 2020 Mar 5;6(1):16. doi: 10.1038/s41572-020-0151-7. PMID 32139695
- [Background] Coles AH, Tisminetzky M, Yarzebski J, Lessard D, Gore JM, Darling CE, Goldberg RJ. Magnitude of and Prognostic Factors Associated With 1-Year Mortality After Hospital Discharge for Acute Decompensated Heart Failure Based on Ejection Fraction Findings. J Am Heart Assoc. 2015 Dec 23;4(12):e002303. doi: 10.1161/JAHA.115.002303. PMID 26702084
- [Background] Di Tano G, De Maria R, Gonzini L, Aspromonte N, Di Lenarda A, Feola M, Marini M, Milli M, Misuraca G, Mortara A, Oliva F, Pulignano G, Russo G, Senni M, Tavazzi L; IN-HF Outcome Investigators. The 30-day metric in acute heart failure revisited: data from IN-HF Outcome, an Italian nationwide cardiology registry. Eur J Heart Fail. 2015 Oct;17(10):1032-41. doi: 10.1002/ejhf.290. Epub 2015 May 27. PMID 26018852
- [Background] Wang H, Chai K, Du M, Wang S, Cai JP, Li Y, Zeng P, Zhu W, Zhan S, Yang J. Prevalence and Incidence of Heart Failure Among Urban Patients in China: A National Population-Based Analysis. Circ Heart Fail. 2021 Oct;14(10):e008406. doi: 10.1161/CIRCHEARTFAILURE.121.008406. Epub 2021 Aug 28. PMID 34455858
- [Background] McLean RR, Kiel DP. Developing consensus criteria for sarcopenia: an update. J Bone Miner Res. 2015 Apr;30(4):588-92. doi: 10.1002/jbmr.2492. PMID 25735999
- [Background] Kalafateli M, Mantzoukis K, Choi Yau Y, Mohammad AO, Arora S, Rodrigues S, de Vos M, Papadimitriou K, Thorburn D, O'Beirne J, Patch D, Pinzani M, Morgan MY, Agarwal B, Yu D, Burroughs AK, Tsochatzis EA. Malnutrition and sarcopenia predict post-liver transplantation outcomes independently of the Model for End-stage Liver Disease score. J Cachexia Sarcopenia Muscle. 2017 Feb;8(1):113-121. doi: 10.1002/jcsm.12095. Epub 2016 Feb 1. PMID 27239424
- [Background] Chen R, Xu J, Wang Y, Jiang B, Xu X, Lan Y, Wang J, Lin X. Prevalence of sarcopenia and its association with clinical outcomes in heart failure: An updated meta-analysis and systematic review. Clin Cardiol. 2023 Mar;46(3):260-268. doi: 10.1002/clc.23970. Epub 2023 Jan 16. PMID 36644878
- [Background] von Haehling S, Garfias Macedo T, Valentova M, Anker MS, Ebner N, Bekfani T, Haarmann H, Schefold JC, Lainscak M, Cleland JGF, Doehner W, Hasenfuss G, Anker SD. Muscle wasting as an independent predictor of survival in patients with chronic heart failure. J Cachexia Sarcopenia Muscle. 2020 Oct;11(5):1242-1249. doi: 10.1002/jcsm.12603. Epub 2020 Aug 6. PMID 32767518
- [Background] Curcio F, Testa G, Liguori I, Papillo M, Flocco V, Panicara V, Galizia G, Della-Morte D, Gargiulo G, Cacciatore F, Bonaduce D, Landi F, Abete P. Sarcopenia and Heart Failure. Nutrients. 2020 Jan 14;12(1):211. doi: 10.3390/nu12010211. PMID 31947528
- [Background] Yin J, Lu X, Qian Z, Xu W, Zhou X. New insights into the pathogenesis and treatment of sarcopenia in chronic heart failure. Theranostics. 2019 May 31;9(14):4019-4029. doi: 10.7150/thno.33000. eCollection 2019. PMID 31281529
- [Background] Eschalier R, Massoullie G, Boirie Y, Blanquet M, Mulliez A, Tartiere PL, Anker S, D'Agrosa Boiteux MC, Richard R, Jean F, Combaret N, Souteyrand G, Riocreux C, Pereira B, Motreff P, Stolt P, Rossignol P, Clerfond G. Sarcopenia in patients after an episode of acute decompensated heart failure: An underdiagnosed problem with serious impact. Clin Nutr. 2021 Jun;40(6):4490-4499. doi: 10.1016/j.clnu.2020.12.033. Epub 2021 Jan 9. PMID 33483182
- [Background] Matsumura K, Teranaka W, Matsumoto H, Fujii K, Tsujimoto S, Otagaki M, Morishita S, Hashimoto K, Shibutani H, Yamamoto Y, Shiojima I. Loss of skeletal muscle mass predicts cardiac death in heart failure with a preserved ejection fraction but not heart failure with a reduced ejection fraction. ESC Heart Fail. 2020 Dec;7(6):4100-4107. doi: 10.1002/ehf2.13021. Epub 2020 Sep 23. PMID 32964678
- [Background] Lopez PD, Nepal P, Akinlonu A, Nekkalapudi D, Kim K, Cativo EH, Visco F, Mushiyev S, Pekler G. Low Skeletal Muscle Mass Independently Predicts Mortality in Patients with Chronic Heart Failure after an Acute Hospitalization. Cardiology. 2019;142(1):28-36. doi: 10.1159/000496460. Epub 2019 Mar 20. PMID 30893691
- [Background] Liu C, Cheng KY, Tong X, Cheung WH, Chow SK, Law SW, Wong RMY. The role of obesity in sarcopenia and the optimal body composition to prevent against sarcopenia and obesity. Front Endocrinol (Lausanne). 2023 Mar 1;14:1077255. doi: 10.3389/fendo.2023.1077255. eCollection 2023. PMID 36936175
- [Background] Shibasaki K, Ogawa S, Yamada S, Iijima K, Eto M, Kozaki K, Toba K, Ouchi Y, Akishita M. Favorable effect of sympathetic nervous activity on rehabilitation outcomes in frail elderly. J Am Med Dir Assoc. 2015 Sep 1;16(9):799.e7-799.e12. doi: 10.1016/j.jamda.2015.06.007. Epub 2015 Jul 10. PMID 26170032
- [Background] Crawford MH, Bernstein SJ, Deedwania PC, DiMarco JP, Ferrick KJ, Garson A Jr, Green LA, Greene HL, Silka MJ, Stone PH, Tracy CM, Gibbons RJ, Alpert JS, Eagle KA, Gardner TJ, Gregoratos G, Russell RO, Ryan TH, Smith SC Jr. ACC/AHA Guidelines for Ambulatory Electrocardiography. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Revise the Guidelines for Ambulatory Electrocardiography). Developed in collaboration with the North American Society for Pacing and Electrophysiology. J Am Coll Cardiol. 1999 Sep;34(3):912-48. doi: 10.1016/s0735-1097(99)00354-x. No abstract available. PMID 10483977
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Xu ZY, Gao DF, Xu K, Zhou ZQ, Guo YK. The Effect of Posture on Maximum Grip Strength Measurements. J Clin Densitom. 2021 Oct-Dec;24(4):638-644. doi: 10.1016/j.jocd.2021.01.005. Epub 2021 Jan 19. PMID 33526316
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] Green CP, Porter CB, Bresnahan DR, Spertus JA. Development and evaluation of the Kansas City Cardiomyopathy Questionnaire: a new health status measure for heart failure. J Am Coll Cardiol. 2000 Apr;35(5):1245-55. doi: 10.1016/s0735-1097(00)00531-3. PMID 10758967
- [Background] Greene SJ, Butler J, Spertus JA, Hellkamp AS, Vaduganathan M, DeVore AD, Albert NM, Duffy CI, Patterson JH, Thomas L, Williams FB, Hernandez AF, Fonarow GC. Comparison of New York Heart Association Class and Patient-Reported Outcomes for Heart Failure With Reduced Ejection Fraction. JAMA Cardiol. 2021 May 1;6(5):522-531. doi: 10.1001/jamacardio.2021.0372. PMID 33760037
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Cooper LB, Mentz RJ, Sun JL, Schulte PJ, Fleg JL, Cooper LS, Pina IL, Leifer ES, Kraus WE, Whellan DJ, Keteyian SJ, O'Connor CM. Psychosocial Factors, Exercise Adherence, and Outcomes in Heart Failure Patients: Insights From Heart Failure: A Controlled Trial Investigating Outcomes of Exercise Training (HF-ACTION). Circ Heart Fail. 2015 Nov;8(6):1044-51. doi: 10.1161/CIRCHEARTFAILURE.115.002327. PMID 26578668
- [Background] Maeda D, Matsue Y, Kagiyama N, Jujo K, Saito K, Kamiya K, Saito H, Ogasahara Y, Maekawa E, Konishi M, Kitai T, Iwata K, Wada H, Hiki M, Dotare T, Sunayama T, Kasai T, Nagamatsu H, Ozawa T, Izawa K, Yamamoto S, Aizawa N, Wakaume K, Oka K, Momomura SI, Minamino T. Sex differences in the prevalence and prognostic impact of physical frailty and sarcopenia among older patients with heart failure. Nutr Metab Cardiovasc Dis. 2022 Feb;32(2):365-372. doi: 10.1016/j.numecd.2021.10.012. Epub 2021 Oct 23. PMID 34893406
- [Background] McNallan SM, Chamberlain AM, Gerber Y, Singh M, Kane RL, Weston SA, Dunlay SM, Jiang R, Roger VL. Measuring frailty in heart failure: a community perspective. Am Heart J. 2013 Oct;166(4):768-74. doi: 10.1016/j.ahj.2013.07.008. Epub 2013 Sep 17. PMID 24093859
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Shah SJ, Cowie MR, Wachter R, Szecsody P, Shi V, Ibram G, Hu M, Zhao Z, Gong J, Pieske B. Baseline characteristics of patients in the PARALLAX trial: insights into quality of life and exercise capacity in heart failure with preserved ejection fraction. Eur J Heart Fail. 2021 Sep;23(9):1541-1551. doi: 10.1002/ejhf.2277. Epub 2021 Jul 26. PMID 34170062
- [Background] Allen LA, Gheorghiade M, Reid KJ, Dunlay SM, Chan PS, Hauptman PJ, Zannad F, Konstam MA, Spertus JA. Identifying patients hospitalized with heart failure at risk for unfavorable future quality of life. Circ Cardiovasc Qual Outcomes. 2011 Jul;4(4):389-98. doi: 10.1161/CIRCOUTCOMES.110.958009. Epub 2011 Jun 21. PMID 21693723
- [Background] Konishi M, Kagiyama N, Kamiya K, Saito H, Saito K, Ogasahara Y, Maekawa E, Misumi T, Kitai T, Iwata K, Jujo K, Wada H, Kasai T, Nagamatsu H, Ozawa T, Izawa K, Yamamoto S, Aizawa N, Makino A, Oka K, Momomura SI, Matsue Y. Impact of sarcopenia on prognosis in patients with heart failure with reduced and preserved ejection fraction. Eur J Prev Cardiol. 2021 Aug 9;28(9):1022-1029. doi: 10.1093/eurjpc/zwaa117. PMID 33624112
- [Background] Sayer AA, Cruz-Jentoft A. Sarcopenia definition, diagnosis and treatment: consensus is growing. Age Ageing. 2022 Oct 6;51(10):afac220. doi: 10.1093/ageing/afac220. PMID 36273495
- [Background] Kono Y, Izawa H, Aoyagi Y, Ishikawa A, Sugiura T, Mori E, Ueda S, Fujiwara W, Hayashi M, Saitoh E. The difference in determinant factor of six-minute walking distance between sarcopenic and non-sarcopenic elderly patients with heart failure. J Cardiol. 2020 Jan;75(1):42-46. doi: 10.1016/j.jjcc.2019.07.002. Epub 2019 Aug 4. PMID 31387751
- [Background] Zhang Y, Zhang J, Ni W, Yuan X, Zhang H, Li P, Xu J, Zhao Z. Sarcopenia in heart failure: a systematic review and meta-analysis. ESC Heart Fail. 2021 Apr;8(2):1007-1017. doi: 10.1002/ehf2.13255. Epub 2021 Feb 11. PMID 33576177
- [Background] Del Buono MG, Arena R, Borlaug BA, Carbone S, Canada JM, Kirkman DL, Garten R, Rodriguez-Miguelez P, Guazzi M, Lavie CJ, Abbate A. Exercise Intolerance in Patients With Heart Failure: JACC State-of-the-Art Review. J Am Coll Cardiol. 2019 May 7;73(17):2209-2225. doi: 10.1016/j.jacc.2019.01.072. PMID 31047010
- [Background] Damluji AA, Alfaraidhy M, AlHajri N, Rohant NN, Kumar M, Al Malouf C, Bahrainy S, Ji Kwak M, Batchelor WB, Forman DE, Rich MW, Kirkpatrick J, Krishnaswami A, Alexander KP, Gerstenblith G, Cawthon P, deFilippi CR, Goyal P. Sarcopenia and Cardiovascular Diseases. Circulation. 2023 May 16;147(20):1534-1553. doi: 10.1161/CIRCULATIONAHA.123.064071. Epub 2023 May 15. PMID 37186680
- [Background] Geraci A, Calvani R, Ferri E, Marzetti E, Arosio B, Cesari M. Sarcopenia and Menopause: The Role of Estradiol. Front Endocrinol (Lausanne). 2021 May 19;12:682012. doi: 10.3389/fendo.2021.682012. eCollection 2021. PMID 34093446
- [Background] Dauriz M, Mantovani A, Bonapace S, Verlato G, Zoppini G, Bonora E, Targher G. Prognostic Impact of Diabetes on Long-term Survival Outcomes in Patients With Heart Failure: A Meta-analysis. Diabetes Care. 2017 Nov;40(11):1597-1605. doi: 10.2337/dc17-0697. PMID 29061587
- [Background] Mentz RJ, Kelly JP, von Lueder TG, Voors AA, Lam CS, Cowie MR, Kjeldsen K, Jankowska EA, Atar D, Butler J, Fiuzat M, Zannad F, Pitt B, O'Connor CM. Noncardiac comorbidities in heart failure with reduced versus preserved ejection fraction. J Am Coll Cardiol. 2014 Dec 2;64(21):2281-93. doi: 10.1016/j.jacc.2014.08.036. Epub 2014 Nov 24. PMID 25456761
- [Background] Ghio S, Mercurio V, Attanasio A, Asile G, Tocchetti CG, Paolillo S. Prognostic impact of diabetes in chronic and acute heart failure. Heart Fail Rev. 2023 May;28(3):577-583. doi: 10.1007/s10741-021-10193-8. Epub 2021 Nov 22. PMID 34811630
- [Background] Anker SD, Ponikowski P, Varney S, Chua TP, Clark AL, Webb-Peploe KM, Harrington D, Kox WJ, Poole-Wilson PA, Coats AJ. Wasting as independent risk factor for mortality in chronic heart failure. Lancet. 1997 Apr 12;349(9058):1050-3. doi: 10.1016/S0140-6736(96)07015-8. PMID 9107242
- [Background] Niedziela JT, Hudzik B, Strojek K, Polonski L, Gasior M, Rozentryt P. Weight loss in heart failure is associated with increased mortality only in non-obese patients without diabetes. J Cachexia Sarcopenia Muscle. 2019 Dec;10(6):1307-1315. doi: 10.1002/jcsm.12471. Epub 2019 Aug 9. PMID 31397095
- [Derived] Bai B, Li D, Xu M, Liao Y, Zhou H, Liu F, Li W, Ma H. Clinical implication of sarcopenia in patients with acute decompensated heart failure: Design and rationale. ESC Heart Fail. 2025 Feb;12(1):640-648. doi: 10.1002/ehf2.15044. Epub 2024 Sep 3. PMID 39225327